CLINICAL TRIAL: NCT00117455
Title: A Randomised, Multi-Centre, Double-Blind Study of Peripheral Blood Progenitor Cell (PBPC) Mobilisation by Chemotherapy With Pegfilgrastim or Filgrastim for Autologous Transplantation in Subjects With Non-Hodgkin's Lymphoma
Brief Title: A Study of Peripheral Blood Progenitor Cell (PBPC) Mobilisation by Chemotherapy With Pegfilgrastim or Filgrastim in Subjects With Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20020113
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Last update posted 2008-05-16 (Estimated); Status verified 2008-05

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: ICE; BEAM; PBPC transplant
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — pegfilgrastim; Filgrastim

INTERVENTIONS:
Drug: pegfilgrastim
Drug: filgrastim

SUMMARY:
The purpose of this study is to evaluate the ability of two different fixed doses of pegfilgrastim (6mg and 12mg) and a by-weight dose of filgrastim (5ug/kg/day) for the mobilisation and collection of PBPCs for autologous transplantation after chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Subjects with non-Hodgkin's lymphoma (NHL) who are considered to be suitable candidates for autologous PBPC transplantation per institution guidelines - ECOG 0-2 inclusive - ANC greater than 1.5 x 10^9/L; PLT greater than 100 x 10^9/L Exclusion Criteria: - More than one line (regimen) of previous chemotherapy treatment and more than 2 cycles of any premobilisation salvage chemotherapy prior to enrolment. Patients were also to be excluded from the study if they had received any salvage chemotherapy containing the following agents: procarbazine, nitrogen mustard, nitrosoureas (including BCNU), melphalan and fludarabine. - Previous bone marrow or PBPC transplant - Greater than 20% bone marrow involvement of the disease at time of screening, as demonstrated by biopsy - Prior total nodal irradiation or any radiotherapy in the past 4 weeks - Serum creatinine greater than 1.5 x upper limit of institutional normal range - Total serum bilirubin greater than 2 x upper limit of institutional normal range - Current diagnosis of splenomegaly not related to lymphoma - History of prior malignancy, except for lymphoma, curatively treated basal cell carcinoma, squamous cell carcinoma, in-situ cervical carcinoma or a surgically cured malignancy - Any premalignant myeloid condition or any malignancy with myeloid characteristics (e.g., myelodysplastic syndromes, acute or chronic myelogenous leukaemia) - Significant non-malignant disease, including documented HIV infection, uncontrolled hypertension (diastolic blood pressure greater than 115 mmHg), unstable angina, congestive heart failure (greater than NY Heart Association Class II), poorly controlled diabetes, coronary angioplasty within 6 months, uncontrolled atrial or ventricular cardiac arrhythmias, or active hepatitis C - Haematopoietic growth factors administered within 1 week of study entry. If growth factor support was given during previous chemotherapy cycles, WBC less than 15.0 x 10^9/L was required at enrolment - Treatment with Interferon® during the last 3 months - Known hypersensitivity to E. coli-derived pharmaceutical products (e.g., filgrastim, HUMULIN® insulin, L-asparaginase) - Subject had previously been randomised into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Adequate collection of PBPC's to enable transplant following high dose chemotherapy

SECONDARY OUTCOMES:
Time to engraftment post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Russell N, Mesters R, Schubert J, Boogaerts M, Johnsen HE, Canizo CD, Baker N, Barker P, Skacel T, Schmitz N. A phase 2 pilot study of pegfilgrastim and filgrastim for mobilizing peripheral blood progenitor cells in patients with non-Hodgkin's lymphoma receiving chemotherapy. Haematologica. 2008 Mar;93(3):405-12. doi: 10.3324/haematol.11287. Epub 2008 Feb 11. PMID 18268285
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf